CLINICAL TRIAL: NCT03997474
Title: An Open-Label, Multi-Centre Phase I/IIa Study Evaluating the Safety and Clinical Activity of Neoantigen Reactive T Cells in Patients With Metastatic or Recurrent Melanoma
Brief Title: ATL001 in Patients With Metastatic or Recurrent Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Achilles Therapeutics UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATX-ME-001
Record Dates: First submitted 2019-02-04; First posted 2019-06-25 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Following lymphodepletion, infusion of cell therapy product ATL001, followed by a low dose regimen of IL- 2.
  Interventions: Biological: ATL001
- Cohort B (Experimental): Following lymphodepletion, infusion of cell therapy product ATL001 in combination with a checkpoint inhibitor, followed by a low dose regimen of IL-2.
  Interventions: Biological: ATL001; Drug: Checkpoint Inhibitor
- Cohort C (Experimental): Following lymphodepletion, infusion of cell therapy product ATL001, followed by a higher dose regimen of IL-2.
  Interventions: Biological: ATL001

INTERVENTIONS:
Biological: ATL001 — ATL001 infusion
Drug: Checkpoint Inhibitor — Nivolumab
  Arms: Cohort B

SUMMARY:
This is a first-in-human, open-label, multi-centre, phase I/IIa study to characterize the safety and clinical activity of ATL001, autologous clonal neoantigen reactive T cells (cNeT) administered intravenously in adults with metastatic or recurrent melanoma.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multi-centre, phase I/IIa study to characterize the safety and clinical activity autologous clonal neoantigen reactive T cells (cNeT) administered intravenously in adults with metastatic or recurrent melanoma.

Patients will initially enter the study for procurement of tumour materials required to manufacture ATL001.Following manufacture of ATL001, the product will be given back to eligible patients following lymphodepletion.

Patients will be followed up for a period of 24 months post ATL001 infusion in the study.

Patients will continue to be followed up for a minimum of 5 years, as part of a separate Long Term Follow Up Protocol, or, if the separate protocol is not available at the study site, within this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old.
2. Patient must have given written informed consent.
3. Patients must have histologically confirmed diagnosis of melanoma.
4. Patient is considered medically fit to undergo procurement of starting material and ATL001 administration procedures.
5. ECOG Performance Status 0-1.
6. Adequate organ function per the laboratory parameters defined in the protocol.
7. Female patients who are of childbearing potential must agree to use a highly effective method of contraception during the study for at least 12 months after the ATL001 infusion. Non-sterilised male participants who intend to be sexually active with a female partner of childbearing potential must use an acceptable method of contraception from the time of screening, throughout the duration of the study and for at least 6 months after the ATL001 infusion.
8. Anticipated life expectancy ≥ 6 months at the time of tissue procurement.
9. Measurable disease according to RECIST v1.1 criteria. Additional inclusion criteria will apply as per the study protocol.

Exclusion Criteria:

1. Patients with known leptomeningeal disease or untreated, symptomatic or progressing central nervous system (CNS) metastases. Lesions should be clinically and radiologically stable for 2 months after treatment and should not require steroids.
2. Patients with ocular, acral or mucosal melanoma.
3. Patients with hepatitis B or C, human immunodeficiency virus infection (HIV 1/2), syphilis or HTLV I/II infection.
4. Patients requiring immunosuppressive treatments.
5. Patients requiring regular steroids at a dose higher than prednisolone 10mg/day (or equivalent).
6. Patients with clinically significant, progressive, and/or uncontrolled renal, hepatic, haematological, endocrine, pulmonary, cardiac, gastroenterological, or neurological disease.
7. Patients with a history of immune mediated (CNS) toxicity or ≥ Grade 2 diarrhoea/colitis caused by, , previous immunotherapy within the past 6 months.
8. Patients who are pregnant or breastfeeding.
9. Patients who have undergone major surgery in the previous 3 weeks.
10. Patients with an active concurrent cancer or a history of cancer within the past 3 years (except for in situ carcinomas, early prostate cancer with normal Prostate-Specific Antigen (PSA) or non-melanomatous skin cancers).
11. Patients with a history of organ transplantation.
12. Patients who have previously received any investigational cell or gene therapies.
13. Patients with contraindications for protocol specified agents.

Additional Exclusion criteria will apply as per the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Achilles Therapeutics UK Limited
Locations (10):
- Spain (2):
  - Instituto de Investigación Sanitaria Fundación Jimenez Díaz, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC) Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge
  - University College London Hospitals (UCLH) NHS Foundation Trust, University College Hospital, London
  - Royal Free London NHS Foundation Trust, Royal Free Hospital, London
  - Guys and St Thomas' NHS Foundation Trust, Guy's Hospital, London
  - The Royal Marsden NHS Foundation Trust, The Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Christie Hospital, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 9 | 2 | 2
Completed | 0 | 0 | 0
Not Completed | 9 | 2 | 2
Not completed — Death | 6 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — study terminated by sponsor | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No differences.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 9 | 2 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 2 | 12
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.49) | 59.5 (4.95) | 36.5 (4.95) | 49.7 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 4
  Male | 7 | 2 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 2 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 2 | 2 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 2 | 1 | 12
  Spain | 0 | 0 | 1 | 1
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.52 (4.922) | 25.55 (2.052) | 22.90 (1.838) | 27.2 (4.651)
Baseline ECOG performance status [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) performance score is a widely used scale to assess a patient's level of functioning, particularly in cancer clinical trials.
  This assessment was performed at the Baseline Screening period by the clinical research teams when they reviewed their patients.
  Score 0: Fully active, able to carry out all pre-disease performance without restrictions.
  Score 1: Restricted in physically strenuous activity but ambulatory and able to perform light work.
  Participants
    Grade 0 | 2 | 1 | 1 | 4
    Grade 1 | 7 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Treatment Emergent Adverse Events to Evaluate Safety and Tolerability: CTCAE
Description: Evaluate treatment-emergent adverse events (TEAEs) and serious AEs, per CTCAE, by incidence, severity and relationship to ATL001
Time Frame: 60 months due to early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 9 | 2 | 2
Participants
  TEAEs | 9 | 2 | 2
  TEAEs related to any component of study treatment | 8 | 2 | 2
  Lymphodepletion related TEAEs | 8 | 1 | 2
  ATL001 related TEAEs IL-2 related TEAEs Serious TEAEs | 5 | 2 | 2
  IL-2 related TEAEs | 7 | 2 | 2
  Nivolumab related TEAEs | 0 | 0 | 0
  Serious TEAEs | 3 | 1 | 0
  Serious TEAEs related to any component of study treatment | 1 | 1 | 0
  Serious Lymphodepletion related TEAEs | 0 | 0 | 0
  Serious ATL001 related TEAEs | 1 | 1 | 0
  Serious IL-2 related TEAEs | 1 | 1 | 0
  Serious Nivolumab related TEAEs | 0 | 0 | 0
  TEAEs with CTCAE grade >= 3 | 6 | 2 | 1
  TEAEs with CTCAE grade >= 3 related to any component of study treatment | 5 | 2 | 1
  Lymphodepletion related TEAEs with CTCAE grade >= 3 | 4 | 1 | 1
  ATL001 related TEAEs with CTCAE grade >= 3 | 2 | 1 | 0
  IL-2 related TEAEs with CTCAE grade >= 3 | 2 | 2 | 0
  Nivolumab related TEAEs with CTCAE grade >= 3 | 0 | 1 | 0
  TEAEs leading to death | 0 | 1 | 0
  TEAEs leading to death related to any component of study treatment | 0 | 0 | 0
  SAEs | 3 | 2 | 1

2. Secondary Outcome: Disease Assessment for Change From Baseline in Tumour Size
Description: Evaluate the clinical activity of ATL001 in patients with recurrent or metastatic melanoma using change from baseline in tumour size at week 6, week 12 and best overall change from baseline, as assessed by investigator and independent central review (ICR).
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

3. Secondary Outcome: Disease Assessment for Overall Response Rate
Description: Evaluate the endpoint of overall response rate (ORR), as assessed by investigator and ICR, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and immune modified RECIST( im-RECIST).
  RECIST v1.1 (Response Evaluation Criteria in Solid Tumors) is a standardized system for measuring tumor response to treatment in clinical trials. Tumors are assessed by imaging (e.g., CT or MRI) based on changes in size. Responses are categorized as:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): ≥30% reduction in the sum of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD).
  Progressive Disease (PD): ≥20% increase in the sum of target lesions, or appearance of new lesions.
  These criteria help assess the efficacy of treatments in solid tumors supported by im-RECIST in immunotherapy.
Time Frame: Every 6 weeks for 6 months, then every 3 months (up to 60 months due to early study termination)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 9 | 2 | 2
Participants
  Responders | 0 | 0 | 0
  Non-Responders | 9 | 2 | 2

4. Secondary Outcome: Disease Assessment for Time to Response and Duration of Response
Description: Evaluate the endpoints of time to response and duration of response (DOR) by the investigator and ICR, per RECIST v1.1 and im-RECIST.
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

5. Secondary Outcome: Disease Assessment for Disease Control Rate
Description: Evaluate the endpoints of disease control rate (DCR) as assessed by the investigator and ICR per RECIST v1.1 and im-RECIST.
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

6. Secondary Outcome: Disease Assessment for Progression-Free Survival
Description: Evaluate the efficacy endpoints of progression-free survival (PFS) as assessed by the investigator and ICR per RECIST v1.1 and im-RECIST.
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Description: Evaluate overall survival (OS) by investigator
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each patient that received ATL001 would have been followed up for 24 months, to withdrawal of consent or death. Patients would then continue to be followed up for a minimum of 5 years as part of long term follow up. The study was terminated early due to sponsor decision. The Median follow-up period was 12 weeks (range: 3 - 48 weeks).
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 8/9 | 2/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=9) | Cohort B (N=2) | Cohort C (N=2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drain site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=9) | Cohort B (N=2) | Cohort C (N=2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (3)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 2 (5) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (6) | 1 (3) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 4 (5) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (12) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 1 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Euthyroid sick syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 2 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (5) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (5) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 2 (6) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (5) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (5) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (6) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Intention tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gram stain positive (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Range of other disclosure agreements across study sites. Following multi-center publication of the Study results made by Sponsor, the Institution and/or Principal Investigator may publish data or results from the Study provided the Sponsor is given 45 to 90 days to review and/or make comments and suggestions where pertinent.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03997474/Prot_SAP_000.pdf